CLINICAL TRIAL: NCT06372223
Title: A Single-center, Randomized, Open, Single-dose, Two-cycle, Two-sequence Crossover Food Effect Study of SPH5030 Tablets in Healthy Chinese Adult Subjects.
Brief Title: A Food Effect Study of SPH5030 Tablets.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPH5030-102
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: SPH5030
- Group B (Experimental)
  Interventions: Drug: SPH5030

INTERVENTIONS:
Drug: SPH5030 — SPH5030 tablets：400mg,orally, Dosing in the fasted state followed by fed dosing.
  Arms: Group A
Drug: SPH5030 — SPH5030 tablets：400mg, orally, Dosing in the fed state followed by fasted dosing.
  Arms: Group B

SUMMARY:
The purpose of this study is to evaluate the food effect of SPH5030 tablets in healthy Chinese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed subjects who voluntarily sign the ICF；
2. Females who are not pregnant, non-lactating. Subjects who complied with the contraceptive requirements of the protocol.

Exclusion Criteria:

1. Subjects with any medical history assessed by the investigator that unsuitable for participation in a clinical study;
2. Subjects with abnormal test results during the screening period；
3. Subjects who have difficulty in venous blood collection;
4. Subjects who cannot accept uniform diet or have difficulty swallowing;
5. Other situations that meet the exclusion criteria.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Approximately 2 months
  PK（Pharmacokinetics）
Peak time（Tmax） | Approximately 2 months
  PK（Pharmacokinetics）
Area under the plasma concentration versus time curve (AUC) | Approximately 2 months
  PK（Pharmacokinetics）

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Approximately 2 months
  Adverse event type, incidence, duration

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second Hospital ,Sichuan University, Chengdu, China